CLINICAL TRIAL: NCT04560725
Title: PSMA Specific [68Ga]-P137 Peptide Probe for PET Imaging in Prostate Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Hua Zhu, Associate Professor, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020KT107
Record Dates: First submitted 2020-09-18; First posted 2020-09-23 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Prostate Cancer
Keywords: PSMA
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [68Ga] P137 (Experimental): Imaging cohort. All study participants will be allocated to this arm (single-arm study).Study participants will undergo [68Ga]P137 PET/CT scans.
  Interventions: Drug: 11C-Choline

INTERVENTIONS:
Drug: 11C-Choline — 11C-choline (0.05-0.1mCi/kg) was injected intravenously one week before or after the [68Ga]P137 PET/CT examination, and imaging of the head and body cadres was performed 20 min after the injection using Philips Gemini TF16 or Siemens Biograph M-CT flow PET/CT
  Other Names: 11C-CH

SUMMARY:
To study the radioactive uptake of [68Ga]P137 in the lesion sites of PCa patients and evaluate the ability of [68Ga]P137 to detect PSMA overexpression in PCa patients (especially those with recurrent or advanced PCa).

DETAILED DESCRIPTION:
Prostate cancer is the most common malignancy of the male reproductive system.Prostate specific membrane antigen is a highly specific prostatic epithelial cell membrane antigen, which is highly expressed in solid tumors such as prostate cancer. More than 90% of prostate cancer cells express PSMA, so PSMA can be used as an important imaging target for prostate cancer.Positron emission tomography has the advantages of non-invasive, high resolution and high sensitivity, etc. The PET tracer based on PSMA radiographic label is developing rapidly, which is of great significance for the early diagnosis, prognosis and treatment of prostate cancer.Used for radionuclide 68Ga has a half-life of PET imaging (T1/2 = 68 min) is appropriate, prepared from 68Ge-68Ga generator, relatively low cost, coordination marking method is simple, easy to realize automatic synthesis technology and advantages of medicine preparation, so 68Ga- labeled PSMA targeted molecular probe in prostate cancer has been widely applied in the diagnosis of disease.

[68Ga]P137 is a novel PSMA targeted molecular probe labeled with 68Ga. DOTA is used as a bifunctional linker to coordinate with 68Ga3+. The labeling method is simple, the biological stability is high, the tumor site has obvious radioactive enrichment, and the imaging effect is superior.This project provides research on [68Ga]P137 PET/CT imaging for patients with suspected PCa, and provides basis for early diagnosis of PCa, formulation of treatment plan and efficacy evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Men over 18 years of age need to undergo [68Ga]P137 PET/CT examination for suspected prostate cancer.
* The patients can fully understand and voluntarily participate in this experiment, and sign the informed consent.

Exclusion Criteria:

* Significant hepatic or renal dysfunction;
* Patients with malignant tumors other than prostate cancer within 2 years;
* Ready to pregnant;
* The patient can not tolerate all clinical tests.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-10-22 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
SUV | 2 years
  The uptake of the tracer in the primary and metastatic tumor lesions by measuring standardized uptake value（SUV）on PET/CT

SECONDARY OUTCOMES:
ROC | 2 years
  The curve of the relationship between sensitivity and specificity

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Duan X, Cao Z, Zhu H, Liu C, Zhang X, Zhang J, Ren Y, Liu F, Cai X, Guo X, Xi Z, Pomper MG, Yang Z, Fan Y, Yang X. 68Ga-labeled ODAP-Urea-based PSMA agents in prostate cancer: first-in-human imaging of an optimized agent. Eur J Nucl Med Mol Imaging. 2022 Feb;49(3):1030-1040. doi: 10.1007/s00259-021-05486-x. Epub 2021 Aug 28. PMID 34453203